CLINICAL TRIAL: NCT01500044
Title: Cervical Radiculopathy: A Randomized Clinical Trial Evaluating the Effect of Mobilizations and Exercises Targeting the Opening of Intervertebral Foramens
Brief Title: Effect of Mobilizations and Exercises Targeting the Opening of Intervertebral Foramens Following Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-12-#09
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Radiculopathy
Keywords: Radiculopathy; Rehabilitation; Mobilization; Exercise; Physical Therapy
MeSH Terms: conditions — Radiculopathy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Rehabilitation Program (Active Comparator): The conventional program consists in cervicothoracic mobilizations and stabilization exercises. This program is based on the intervention used in clinical practice, and on programs proposed in two RCTs evaluating individuals with neck and arm pain that do not include any specific mobilization or exercise leading to the opening of the intervertebral foramen. Four mobilisation techniques will be executed at each treatment session. However, the therapists will not be allowed to use techniques that specifically open the intervertebral foramen of the affected segment, two segments above and two segments below.
  Interventions: Procedure: Conventional Rehabilitation Program
- Program targeting the opening of foramen (Experimental): The same interventions as for the conventional rehabilitation program will be applied, except:
  Of the four mobilisation techniques, there will be two mandatory techniques targeting the opening of the intervertebral foramen on the same side and at the same level as the radiculopathy: global contralateral rotation mobilisation and ipsilateral lateral shearing in a flexion position. The therapist, according to the biomechanical evaluation results, will choose the two other mobilisation techniques.
  Interventions: Procedure: Program targeting the opening of foramen

INTERVENTIONS:
Procedure: Program targeting the opening of foramen — Rehabilitation intervention that specifically targets the opening of the intervertebral foramen
  Other Names: Specific manual Therapy, Mobilization, Exercises
  Arms: Program targeting the opening of foramen
Procedure: Conventional Rehabilitation Program — Program used in previous randomized clinical trials in this population
  Other Names: Non specific manual therapy, mobilization and exercises
  Arms: Conventional Rehabilitation Program

SUMMARY:
The primary objective of this randomised clinical trial (RCT) is to compare, in terms of disability and pain, an intervention targeting the opening of intervertebral foramens to a conventional physiotherapy intervention, in patients presenting acute or subacute cervical radiculopathies. Based on biomechanical principles, the investigators hypothesis is that the intervention targeting the opening of intervertebral foramens will be significantly more effective in reducing pain and disability than the conventional physiotherapy intervention.

This study is double-blind RCT that will allow the comparison of patients with a cervical radiculopathy randomly assigned to one of two groups: one group will receive a 4-week rehabilitation program targeting the opening of intervertebral foramen, and the second group will receive a 4-week conventional rehabilitation program. Thirty-six subjects will be recruited from participating medical and physiotherapy clinics in the Quebec City area (Canada) and will be evaluated at baseline, at the end of the program and four weeks following the end of the program. The primary outcome measure will be the validated Neck Disability Index (NDI) questionnaire and other secondary measures will include the QuickDASH questionnaire, a numerical pain rating scale, cervicothoracic mobility and patients' perceived global rating of change.

DETAILED DESCRIPTION:
Cervical radiculopathy is a common form of neck pain and has been shown to lead to severe disability. Clinical rehabilitation approaches for cervical radiculopathies commonly include exercise and manual therapy interventions targeting the opening of intervertebral foramen but evidence regarding their effectiveness is scarce.

This double-blind randomised clinical trial will allow the comparison, in terms of pain and disability, of patients presenting a cervical radiculopathy which will have been randomly assigned to one of the two intervention groups: the first group (n = 18) will receive a 4-week rehabilitation program targeting the opening of intervertebral foramen, the second group (n = 18) will receive a 4-week conventional rehabilitation program. Participants will be evaluated on three separate occasions: at baseline (week 0), at the end of the 4-week program (week 4), and four weeks following the end of the program (week 8).

ELIGIBILITY:
Inclusion Criteria:

* pain, paresthesia or numbness in the upper-limb with cervical or periscapular pain for less than 3 months
* at least one neurological sign (dermatomes, myotomes or reflexes) of an inferior motoneuron lesion to the upper-limb
* positive responses to at least 3 of the 4 following clinical tests: Spurling Test, Upper Limb Tension Test, Cervical Distraction Test, and less than 60o of cervical rotation on the impaired side

Exclusion Criteria:

* prior surgery to the cervicothoracic spine
* bilateral upper-limb symptoms
* signs of superior motoneuron impairments (bilateral paresthesia, hyperreflexia, spasticity)
* cervical spine infiltration in the previous four weeks
* current use of steroidal anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Neck Disability Index at 4 weeks | Week 4

SECONDARY OUTCOMES:
Change from baseline in the Numerical Pain Rating Scale at 4 weeks | Week 4
Change from baseline and week 4 in the Numerical Pain Rating Scale at 8 weeks | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

REFERENCES:
- [Derived] Langevin P, Desmeules F, Lamothe M, Robitaille S, Roy JS. Comparison of 2 manual therapy and exercise protocols for cervical radiculopathy: a randomized clinical trial evaluating short-term effects. J Orthop Sports Phys Ther. 2015 Jan;45(1):4-17. doi: 10.2519/jospt.2015.5211. PMID 25420010
- [Derived] Langevin P, Roy JS, Desmeules F. Cervical radiculopathy: study protocol of a randomised clinical trial evaluating the effect of mobilisations and exercises targeting the opening of intervertebral foramen [NCT01500044]. BMC Musculoskelet Disord. 2012 Jan 31;13:10. doi: 10.1186/1471-2474-13-10. PMID 22293092